CLINICAL TRIAL: NCT01852448
Title: Evaluation of the Enteroinsular Axis in Cystic Fibrosis
Brief Title: Genetics of Insulin and Incretins in Cystic Fibrosis
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 12-009589
Record Dates: First submitted 2013-05-09; First posted 2013-05-13 (Estimated); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with Cystic Fibrosis: Blood or saliva sample collection and medical record review.
  Interventions: Genetic: Blood or Saliva Sample Collection

INTERVENTIONS:
Genetic: Blood or Saliva Sample Collection — A blood or saliva sample will be obtained for genotyping of TCF7L2 and approximately ten other genes implicated in type 2 diabetes.

SUMMARY:
Cystic fibrosis related diabetes (CFRD) is associated with worse CF-relevant outcomes.

The mechanisms underlying CFRD development are not fully understood, but recent evidence suggests Type 2 Diabetes Mellitus (T2DM) mechanisms may be involved and may involve incretins (gut secreted hormones that augment insulin secretion in response to a nutrient load).

This study will examine the prevalence of Genome wide association study (GWAS)-implicated T2DM alleles (including TCF7L2) across the spectrum of glucose abnormalities in CF and will use this information to compare incretin and insulin secretion in non-diabetic children and adults with high risk and low risk alleles.

DETAILED DESCRIPTION:
CFRD is associated with worse nutritional status, greater pulmonary function decline, and increased mortality, highlighting its relevance in CF and arises primarily from compromised insulin secretion--traditionally considered a by-product of pancreatic exocrine tissue damage and fibrosis. Recent developments in the field of diabetes are propelling a re-examination of this basic explanation. Genome-wide association studies have associated genetic variants in TCF7L2, a transcription factor implicated in enteroendocrine function, with increased susceptibility to T2DM and CFRD.

The Objectives of this study are to perform targeted sequencing of TCF7L2 and other GWAS-associated T2DM genes in the pediatric and adult CF populations and then to compare insulin secretory capacity, β-cell sensitivity to glucose, and incretin secretion in non-diabetic CF subjects with high and low-risk alleles.

Phase 1 will include 450-500 subjects (Children age>= 2 years, adolescents, and adults) for TCF7L2 genotype and ten other GWAS-implicated T2DM genes. The distribution of TCF7L2 and other GWAS-implicated T2 DM genes across the spectrum of glucose abnormalities will be described. Phase 1 requires a single blood or saliva sample and review of medical records.

ELIGIBILITY:
Inclusion Criteria

1. Subjects age >2y
2. Diagnosis of Cystic Fibrosis
3. For subjects< 18 years, parental/guardian permission (informed consent) and if appropriate, child assent

Exclusion Criteria 1. Established diagnosis of non-CFRD (cystic fibrosis related diabetes) (e.g T1DM)

.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Cystic Fibrosis age >2 yrs
Sampling Method: Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2013-05; Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Blood sample for DNA to genotype TCF7L2 and about 10 other GWAS-implicated T2DM genes. | 1 day
  To examine the prevalence of GWAS-implicated T2DM alleles (including TCF7L2) across the spectrum of glucose abnormalities in children and adults with CF.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Kelly, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - The Children's Hopsital of Philadelphia, Philadelphia, Pennsylvania
  - The University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No